CLINICAL TRIAL: NCT00076076
Title: The FLASH Study: A Randomized, Controlled Study of Roflumilast 250 mcg and 500 mcg Versus Placebo in Patients With Asthma
Brief Title: The FLASH Study: A Study of Roflumilast Versus Placebo in Patients With Asthma (BY217/M2-023)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY217/M2-023
Record Dates: First submitted 2004-01-13; First posted 2004-01-15 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: Roflumilast; Asthma
MeSH Terms: conditions — Asthma | interventions — Roflumilast

INTERVENTIONS:
Drug: Roflumilast

SUMMARY:
The purpose of this study is to confirm the dose of roflumilast to be used for asthma management by comparing the effects of 250 mcg and 500 mcg oral roflumilast with placebo on pulmonary function and asthma symptoms.

ELIGIBILITY:
Main Inclusion Criteria:

* Diagnosis of persistent chronic bronchial asthma
* Baseline lung function within specified parameters
* No change in asthma treatment during the last 4 weeks prior to start of baseline period
* Stable clinical state
* Except for asthma, in good health
* Non-smokers or ex-smokers

Main Exclusion Criteria:

* Poorly controlled asthma
* Diagnosis of chronic pulmonary disease and/or other relevant lung diseases
* Patients using continuously (more than 3 days per week) > 8 puffs/day rescue medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 822
Dates: Start 2003-12; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
change in lung function.

SECONDARY OUTCOMES:
change in morning PEF
asthma symptom score
rescue medication
time to withdrawal due to worsening asthma.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (41):
- United States (39):
  - ALTANA Pharma, Cities in Alabama, Alabama
  - ALTANA Pharma, Cities in Arizona, Arizona
  - ALTANA Pharma, Cities in Arkansas, Arkansas
  - ALTANA Pharma, Cities in California, California
  - ALTANA Pharma, Cities in Colorado, Colorado
  - ALTANA Pharma, Cities in Connecticut, Connecticut
  - ALTANA Pharma, Cities in Delaware, Delaware
  - ALTANA Pharma, Cities in Florida, Florida
  - ALTANA Pharma, Cities in Georgia, Georgia
  - ALTANA Pharma, Cities in Illinois, Illinois
  - ALTANA Pharma, Cities in Indiana, Indiana
  - ALTANA Pharma, Cities in Kansas, Kansas
  - ALTANA Pharma, Cities in Kentucky, Kentucky
  - ALTANA Pharma, Cities in Louisiana, Louisiana
  - ALTANA Pharma, Cities in Maine, Maine
  - ALTANA Pharma, Cities in Maryland, Maryland
  - ALTANA Pharma, Cities in Massachusetts, Massachusetts
  - ALTANA Pharma, Cities in Michigan, Michigan
  - ALTANA Pharma, Cities in Minnesota, Minnesota
  - ALTANA Pharma, Cities in Missouri, Missouri
  - ALTANA Pharma, Cities in Montana, Montana
  - ALTANA Pharma, Cities in Nebraska, Nebraska
  - ALTANA Pharma, Cities in Nevada, Nevada
  - ALTANA Pharma, Cities in New Jersey, New Jersey
  - ALTANA Pharma, Cities in New York, New York
  - ALTANA Pharma, Cities in North Carolina, North Carolina
  - ALTANA Pharma, Cities in Ohio, Ohio
  - ALTANA Pharma, Cities in Oklahoma, Oklahoma
  - ALTANA Pharma, Cities in Oregon, Oregon
  - ALTANA Pharma, Cities in Pennsylvania, Pennsylvania
  - ALTANA Pharma, Cities in Rhode Island, Rhode Island
  - ALTANA Pharma, Cities in South Carolina, South Carolina
  - ALTANA Pharma, Cities in Tennessee, Tennessee
  - ALTANA Pharma, Cities in Texas, Texas
  - ALTANA Pharma, Cities in Utah, Utah
  - ALTANA Pharma, Cities in Vermont, Vermont
  - ALTANA Pharma, Cities in Virginia, Virginia
  - ALTANA Pharma, Cities in Washington, Washington
  - ALTANA Pharma, Cities in West Virginia, West Virginia
- ALTANA Pharma, Cities in Russia, Russia
- ALTANA Pharma, Cities in the Ukraine, Ukraine

REFERENCES:
- [Derived] Chervinsky P, Meltzer EO, Busse W, Ohta K, Bardin P, Bredenbroker D, Bateman ED. Roflumilast for asthma: Safety findings from a pooled analysis of ten clinical studies. Pulm Pharmacol Ther. 2015 Dec;35 Suppl:S28-34. doi: 10.1016/j.pupt.2015.11.003. Epub 2015 Nov 22. PMID 26612545
- [Derived] Meltzer EO, Chervinsky P, Busse W, Ohta K, Bardin P, Bredenbroker D, Bateman ED. Roflumilast for asthma: Efficacy findings in placebo-controlled studies. Pulm Pharmacol Ther. 2015 Dec;35 Suppl:S20-7. doi: 10.1016/j.pupt.2015.10.006. Epub 2015 Oct 21. PMID 26498386
- See also: BY217-M2-023-RDS-2007-01-23.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4474&filename=BY217-M2-023-RDS-2007-01-23.pdf